CLINICAL TRIAL: NCT04217733
Title: A Comparative Study to Assess Safety and Effectiveness of Ethosuximide and Pentoxifylline in the Treatment of Abdominal Pain Related to Irritable Bowel Syndrome
Brief Title: Ethosuximide and Pentoxifylline in the Treatment of Abdominal Pain Related to Irritable Bowel Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sherief Protocol
Record Dates: First submitted 2019-12-29; First posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — mebeverine; Ethosuximide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mebeverine (Active Comparator): Mebeverine 3 times daily for 3 months
  Interventions: Drug: Mebeverine
- Ethosuximide (Experimental): Ethosuxemide 3 times daily for 3 months
  Interventions: Drug: ethosuximide
- Pentoxyifylline (Experimental): pentoxyifylline 2 times daily for 3 months
  Interventions: Drug: pentoxyifylline

INTERVENTIONS:
Drug: pentoxyifylline — Pentoxyifylline two times daily for 3 months
  Arms: Pentoxyifylline
Drug: Mebeverine — Mebeverine 3 times for 3 months
  Arms: Mebeverine
Drug: ethosuximide — ethosuximide 3 times for 3 months
  Arms: Ethosuximide

SUMMARY:
Ethosuximide and pentoxifylline in the treatment of abdominal pain related to irritable bowel syndrome

DETAILED DESCRIPTION:
Ethosuximide and pentoxifylline in the treatment of abdominal pain related to irritable bowel syndrome: Does this add to current treatment?

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 18 years,

  * Man and Women, Negative pregnancy test and effective contraception,
  * IBS defined by the Rome criteria IV
  * During the previous seven days the inclusion visit, average numeric rating scale (NRS) pain ≥ 4.
  * IBS Treatment stable for 1 month

Exclusion Criteria:

* • Breastfeeding

  * Diabetic patients
  * Significant liver function abnormalities (transaminases> 3N, cholestasis) and moderate renal disease (MDRD <60 ml / min)
  * Addiction to alcohol and / or drugs,
  * Antiepileptic drugs taken (epilepsy or chronic pain)
  * Chronic pain of greater intensity than that related to IBS,
  * Known Allergyto succinimides (ethosuximide, methsuximide, phensuximide) and pentoxifylline.
  * History or current severe depression (hospitalization, long-term antidepressant treatment)
  * Psychotic disorders,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with improved Visual analog scales (VAS) for assessment of pain in IBS | 6 months
  the number of patients with improved Visual analog scales (VAS) for assessment of pain in IBS

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Mahmoud Bahaa El dien, Msc, Principal Investigator — Clinical Pharmacy department; Sahar El-Haggar, Prof, Principal Investigator — Clinical pharmacy Department- Tanta University; Sahar Hegazy, Prof., Principal Investigator — Clinical pharmacy Department- Tanta University; Sherief Abd-Elsalam, Ass. Prof., Principal Investigator — Tropical Medicine Department- Tanta University
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Haggar SM, Hegazy SK, Abd-Elsalam SM, Elkaeed EB, Al-Karmalawy AA, Bahaa MM. A Potential Role of Ethosuximide and Pentoxifylline in Relieving Abdominal Pain in Irritable Bowel Syndrome Patients Treated with Mebeverine: A Randomized, Double-Blind, Placebo-Controlled Trial. J Inflamm Res. 2022 Feb 19;15:1159-1172. doi: 10.2147/JIR.S346608. eCollection 2022. PMID 35221706 (Retraction: PMID 35444453 J Inflamm Res. 2022 Apr 14;15:2381-2382)
- [Derived] El-Haggar SM, Hegazy SK, M Abd-Elsalam S, Bahaa MM. Open-label pilot study of ethosuximide as adjunctive therapy for relieving abdominal pain related to Irritable Bowel Syndrome. J Clin Pharm Ther. 2022 Mar;47(3):306-312. doi: 10.1111/jcpt.13556. Epub 2021 Nov 2. PMID 34726293